CLINICAL TRIAL: NCT06271980
Title: Predicting Long-Term Recurrence-Free and Overall Survival in Early-Onset Colorectal Cancer Survivors
Brief Title: Early-Onset Colorectal Cancer Recurrence
Acronym: ENCORE
Status: Completed | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: IRCCS San Raffaele (Other); Institute of Biomedical Research of Salamanca, Salamanca, Spain (Unknown)
Responsible Party: Sponsor
Other Study IDs: 23228/ENCORE
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer Recurrent; Colorectal Cancer; Colorectal Neoplasms; Colorectal Adenocarcinoma; Colorectal Cancer Stage I; Colorectal Cancer Stage II; Colorectal Cancer Stage III
Keywords: Early-Onset; Young-Onset; Surveillance; micro-RNA; Prediction
MeSH Terms: conditions — Colorectal Neoplasms | interventions — enc protein, Drosophila

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Survivors of early-onset colorectal cancer, with recurrent disease (Training Cohort): Survivors of early-onset colorectal cancer who developed recurrent CRC within 60 months from primary tumor treatment, in the first cohort
  Interventions: Other: ENCORE
- Survivors of early-onset colorectal cancer, with no recurrent disease (Training Cohort): Survivors of early-onset colorectal cancer who did not develop recurrent CRC within 60 months from primary tumor treatment, in the first cohort
  Interventions: Other: ENCORE
- Survivors of early-onset colorectal cancer, with recurrent disease (Validation Cohort): Survivors of early-onset colorectal cancer who developed recurrent CRC within 60 months from primary tumor treatment, in the second, independent, validation cohort
  Interventions: Other: ENCORE
- Survivors of early-onset colorectal cancer, with no recurrent disease (Validation Cohort): Survivors of early-onset colorectal cancer who did not develop recurrent CRC within 60 months from primary tumor treatment, in the second, independent, validation cohort
  Interventions: Other: ENCORE

INTERVENTIONS:
Other: ENCORE — A panel of microRNA, whose expression level is tested in macro-dissected formalin-fixed and paraffin-embedded (FFPE) samples derived from the primary tumor.
  Other Names: ENCORE (Early oNset COlorectal cancer REcurrence)

SUMMARY:
Survivors of early-onset colorectal cancer (diagnosed before age 50) may experience colorectal cancer recurrence several years after curative-intent treatments, but clinical guidelines provide unclear guidance on endoscopic surveillance.

This study aims to predict recurrence-free survival and overall survival, in survivors of early-onset colorectal cancer, using a tumor-based molecular assay based on microRNA (ribonucleic acid)

DETAILED DESCRIPTION:
Colorectal cancer (CRC) once predominantly affected older individuals, but in recent years has witnessed a progressive increase in incidence among young adults. Once rare, early-onset colorectal cancer (EOCRC, that is, a CRC diagnosed before the age of 50) now constitutes 10-15% of all newly diagnosed CRC cases and it stands as the first cause of cancer-related death in young men in the US and the second for young women. In the wake of the increasing incidence, the growing population of EOCRC survivors introduces distinctive clinical challenges.

Patients with EOCRC are hypothesized to possess a more biologically active colorectum, susceptible to malignant transformation both earlier in life and later after primary cancer. Indeed, EOCRC survivors encounter an elevated risk of disease recurrence, a risk that may manifest years after primary treatment. These considerations have prompted a trend toward offering more aggressive therapy or endoscopy surveillance, a practice however not substantiated by evidence yet. Scientific societies have also adopted a cautious stance, recognizing the elevated risk while acknowledging the absence of evidence to substantiate an intensified surveillance protocol, which might constitute overtreatment.

In this research effort, the investigators will leverage machine learning to predict recurrence-free survival (RFS) and overall survival (OS) in patients cured of EOCRC. The research plan will employ three phases:

1. After a systematic discovery phase, based on small RNA sequencing, the investigators will identify a panel of candidate biomarkers.
2. The investigators will then develop an assay based on reverse transcription-quantitative polymerase chain reaction (RT-qPCR) and train a machine-learning model to predict recurrence-free and overall survival outcomes
3. The investigators will independently validate the assay.

This assay is provisionally termed "ENCORE" (Early oNset COlorectal cancer REcurrence) and will be tested for recurrence-free and overall survival outcomes up to ten years after treatment.

At the end of this study, this assay will have been developed and validated to help clinical decision-making by predicting both recurrence-free and overall survival in EOCRC survivors.

ELIGIBILITY:
Inclusion Criteria:

* Stage I, II, or III colorectal cancer (TNM classification, 8th edition) diagnosed before the age of 50
* Received standard diagnostic, staging, and therapeutic procedures as per local guidelines, received stage-specific curative-intent resection (with or without systemic therapy, as appropriate)
* Confirmed cancer-free survivors at the time of study inclusion

Exclusion Criteria:

* Hereditary colorectal cancer syndromes (identified through genetic testing)
* Inflammatory bowel diseases
* Lack of written informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Two independent cohorts of early-onset colorectal cancer survivors (stages I-III)
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Recurrence Free Survival | Up to 120 months
  Time from disease treatment to development of recurrent colorectal cancer

SECONDARY OUTCOMES:
Overall Survival | Up to 120 months
  Time from disease treatment to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Goel, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: No
Data collected for the study will be made available to others, including de-identified participant data, at publication, via a signed data access agreement and at the discretion of the investigators' approval of the proposed use of such data.

REFERENCES:
- [Background] Sinicrope FA. Increasing Incidence of Early-Onset Colorectal Cancer. N Engl J Med. 2022 Apr 21;386(16):1547-1558. doi: 10.1056/NEJMra2200869. No abstract available. PMID 35443109
- [Background] Siegel RL, Wagle NS, Cercek A, Smith RA, Jemal A. Colorectal cancer statistics, 2023. CA Cancer J Clin. 2023 May-Jun;73(3):233-254. doi: 10.3322/caac.21772. Epub 2023 Mar 1. PMID 36856579
- [Background] Siegel RL, Giaquinto AN, Jemal A. Cancer statistics, 2024. CA Cancer J Clin. 2024 Jan-Feb;74(1):12-49. doi: 10.3322/caac.21820. Epub 2024 Jan 17. PMID 38230766
- [Background] Kim TJ, Kim ER, Hong SN, Chang DK, Kim YH. Long-Term Outcome and Prognostic Factors of Sporadic Colorectal Cancer in Young Patients: A Large Institutional-Based Retrospective Study. Medicine (Baltimore). 2016 May;95(19):e3641. doi: 10.1097/MD.0000000000003641. PMID 27175682
- [Background] You YN, Dozois EJ, Boardman LA, Aakre J, Huebner M, Larson DW. Young-onset rectal cancer: presentation, pattern of care and long-term oncologic outcomes compared to a matched older-onset cohort. Ann Surg Oncol. 2011 Sep;18(9):2469-76. doi: 10.1245/s10434-011-1674-7. Epub 2011 Mar 30. PMID 21448750
- [Background] Foppa C, Tamburello S, Maroli A, Carvello M, Poliani L, Laghi L, Malesci A, Montorsi M, Perea J, Spinelli A. Early age of onset is an independent predictor for worse disease-free survival in sporadic rectal cancer patients. A comparative analysis of 980 consecutive patients. Eur J Surg Oncol. 2022 Apr;48(4):857-863. doi: 10.1016/j.ejso.2021.10.021. Epub 2021 Oct 28. PMID 34740480
- [Background] Kim SB, Lee HJ, Park SJ, Hong SP, Cheon JH, Kim WH, Kim TI. Comparison of Colonoscopy Surveillance Outcomes Between Young and Older Colorectal Cancer Patients. J Cancer Prev. 2017 Sep;22(3):159-165. doi: 10.15430/JCP.2017.22.3.159. Epub 2017 Sep 30. PMID 29018780
- [Background] Chen FW, Sundaram V, Chew TA, Ladabaum U. Advanced-Stage Colorectal Cancer in Persons Younger Than 50 Years Not Associated With Longer Duration of Symptoms or Time to Diagnosis. Clin Gastroenterol Hepatol. 2017 May;15(5):728-737.e3. doi: 10.1016/j.cgh.2016.10.038. Epub 2016 Nov 14. PMID 27856366
- [Background] Al Maliki H, Monahan KJ. The diagnostic yield of colonoscopic surveillance following resection of early age onset colorectal cancer. United European Gastroenterol J. 2024 May;12(4):469-476. doi: 10.1002/ueg2.12516. Epub 2024 Jan 3. PMID 38170450
- [Background] Peacock O, Vilar E, Guraieb-Trueba M, Thirumurthi S, Chang GJ, You YN. Clinically Significant Metachronous Colorectal Pathology Detected Among Young-Onset Colorectal Cancer Survivors: Implications for Post-Resection Surveillance Guidelines. Gastroenterology. 2022 Dec;163(6):1682-1684.e2. doi: 10.1053/j.gastro.2022.08.030. Epub 2022 Aug 17. No abstract available. PMID 35987446
- [Background] Zaborowski AM, Murphy B, Creavin B, Rogers AC, Kennelly R, Hanly A, Martin ST, O'Connell PR, Sheahan K, Winter DC. Clinicopathological features and oncological outcomes of patients with young-onset rectal cancer. Br J Surg. 2020 Apr;107(5):606-612. doi: 10.1002/bjs.11526. Epub 2020 Mar 9. PMID 32149397
- [Background] Bouvier AM, Latournerie M, Jooste V, Lepage C, Cottet V, Faivre J. The lifelong risk of metachronous colorectal cancer justifies long-term colonoscopic follow-up. Eur J Cancer. 2008 Mar;44(4):522-7. doi: 10.1016/j.ejca.2008.01.007. Epub 2008 Feb 5. PMID 18255278
- [Background] Monahan KJ, Bradshaw N, Dolwani S, Desouza B, Dunlop MG, East JE, Ilyas M, Kaur A, Lalloo F, Latchford A, Rutter MD, Tomlinson I, Thomas HJW, Hill J; Hereditary CRC guidelines eDelphi consensus group. Guidelines for the management of hereditary colorectal cancer from the British Society of Gastroenterology (BSG)/Association of Coloproctology of Great Britain and Ireland (ACPGBI)/United Kingdom Cancer Genetics Group (UKCGG). Gut. 2020 Mar;69(3):411-444. doi: 10.1136/gutjnl-2019-319915. Epub 2019 Nov 28. PMID 31780574
- [Background] Rutter MD, East J, Rees CJ, Cripps N, Docherty J, Dolwani S, Kaye PV, Monahan KJ, Novelli MR, Plumb A, Saunders BP, Thomas-Gibson S, Tolan DJM, Whyte S, Bonnington S, Scope A, Wong R, Hibbert B, Marsh J, Moores B, Cross A, Sharp L. British Society of Gastroenterology/Association of Coloproctology of Great Britain and Ireland/Public Health England post-polypectomy and post-colorectal cancer resection surveillance guidelines. Gut. 2020 Feb;69(2):201-223. doi: 10.1136/gutjnl-2019-319858. Epub 2019 Nov 27. PMID 31776230
- [Background] Cavestro GM, Mannucci A, Balaguer F, Hampel H, Kupfer SS, Repici A, Sartore-Bianchi A, Seppala TT, Valentini V, Boland CR, Brand RE, Buffart TE, Burke CA, Caccialanza R, Cannizzaro R, Cascinu S, Cercek A, Crosbie EJ, Danese S, Dekker E, Daca-Alvarez M, Deni F, Dominguez-Valentin M, Eng C, Goel A, Guillem JG, Houwen BBSL, Kahi C, Kalady MF, Kastrinos F, Kuhn F, Laghi L, Latchford A, Liska D, Lynch P, Malesci A, Mauri G, Meldolesi E, Moller P, Monahan KJ, Moslein G, Murphy CC, Nass K, Ng K, Oliani C, Papaleo E, Patel SG, Puzzono M, Remo A, Ricciardiello L, Ripamonti CI, Siena S, Singh SK, Stadler ZK, Stanich PP, Syngal S, Turi S, Urso ED, Valle L, Vanni VS, Vilar E, Vitellaro M, You YN, Yurgelun MB, Zuppardo RA, Stoffel EM; Associazione Italiana Familiarita Ereditarieta Tumori; Collaborative Group of the Americas on Inherited Gastrointestinal Cancer; European Hereditary Tumour Group, and the International Society for Gastrointestinal Hereditary Tumours. Delphi Initiative for Early-Onset Colorectal Cancer (DIRECt) International Management Guidelines. Clin Gastroenterol Hepatol. 2023 Mar;21(3):581-603.e33. doi: 10.1016/j.cgh.2022.12.006. Epub 2022 Dec 20. PMID 36549470
- [Background] Jung G, Hernandez-Illan E, Moreira L, Balaguer F, Goel A. Epigenetics of colorectal cancer: biomarker and therapeutic potential. Nat Rev Gastroenterol Hepatol. 2020 Feb;17(2):111-130. doi: 10.1038/s41575-019-0230-y. Epub 2020 Jan 3. PMID 31900466
- [Background] Okugawa Y, Grady WM, Goel A. Epigenetic Alterations in Colorectal Cancer: Emerging Biomarkers. Gastroenterology. 2015 Oct;149(5):1204-1225.e12. doi: 10.1053/j.gastro.2015.07.011. Epub 2015 Jul 26. PMID 26216839
- [Background] Nakamura K, Hernandez G, Sharma GG, Wada Y, Banwait JK, Gonzalez N, Perea J, Balaguer F, Takamaru H, Saito Y, Toiyama Y, Kodera Y, Boland CR, Bujanda L, Quintero E, Goel A. A Liquid Biopsy Signature for the Detection of Patients With Early-Onset Colorectal Cancer. Gastroenterology. 2022 Nov;163(5):1242-1251.e2. doi: 10.1053/j.gastro.2022.06.089. Epub 2022 Jul 16. PMID 35850198
- [Derived] Mannucci A, Hernandez G, Uetake H, Yamada Y, Balaguer F, Baba H, Chen T, Chen J, Boland CR, Cavestro GM, Quintero E, Goel A. Prediction of long-term recurrence-free and overall survival in early-onset colorectal cancer: the ENCORE multi-centre study. NPJ Precis Oncol. 2025 Jun 21;9(1):202. doi: 10.1038/s41698-025-00978-7. PMID 40544180